CLINICAL TRIAL: NCT03424590
Title: Libera Efficacy 2 Cycles at Home Study
Brief Title: Connected Ovulation Test Efficacy Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: SPD Development Company Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: PROTOCOL-0987
Record Dates: First submitted 2018-01-25; First posted 2018-02-07 (Actual); Last update posted 2018-10-19 (Actual); Status verified 2018-07

CONDITIONS: Pregnancy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- COTS (Active Comparator): Volunteers will be provided with Clearblue connected Ovulation test system to use during the study period, accortding to the instructions for use.
  Interventions: Device: Clearblue Connected Ovulation Test System
- Control (No Intervention): Volunteers will not be provided with Clearblue Connected Ovulation Test System and will be instructed not to use any other ovulation predictions tests during the study period.

INTERVENTIONS:
Device: Clearblue Connected Ovulation Test System — Urinary LH test to predict ovulation
  Arms: COTS

SUMMARY:
Clearblue Connected Ovulation Test System (COTS) has been designed for home use by women who are either planning or trying for a pregnancy. This study will determine the difference in pregnancy rate of female volunteers seeking to get pregnant who use COTS in comparison to those not using an ovulation product to assist with conception.

ELIGIBILITY:
Inclusion Criteria:

* Actively trying to conceive
* At least 2 regular consecutive cycles since last pregnancy/ miscarriage/ or since stopping breastfeeding
* Willing to use their own smartphone for the duration of this study and to download and install the study app
* Willing to disclose their pregnancy status and provide urine samples to test markers related to pregnancy and fertility
* Have internet access on their phone for the duration of the study
* Willing to give informed consent and comply with the investigational procedures

Exclusion Criteria:

* Currently or previously employed by SPD, Alere, Abbott, Unipath or P&G, or affiliates
* Has an immediate relative* currently or previously employed by SPD, Alere, Abbott, Unipath or P&G or affiliates
* There is a reason why the volunteer should not get pregnant e.g. they are taking a medication or have a medical condition which means they should not get pregnant
* Trying to conceive for more than 6 months (if less than 35 years old) and more than 3 months (if 35 years old or over)
* Has been diagnosed with Polycystic Ovarian Syndrome (PCOS)
* Has PCOS symptoms: very irregular cycles, hirsutism
* Using or has previously used infertility medications or hormone replacement therapy containing hCG or LH (e.g Pregnyl)
* Are taking clomiphene citrate or other ovulation induction drugs
* Using any treatment which may affect the menstrual cycle (e.g. the contraceptive pill)
* Currently pregnant or breastfeeding
* Peri- or post-menopausal, e.g. experiencing symptoms: Irregular menstrual periods, hot flushes, night sweats, sleep disturbances, and mood swings
* Have abnormal liver or kidney function
* Taking medication containing tetracycline
* Using or undergoing any other medical treatment for fertility such as ovulation drugs, artificial insemination and assisted fertility such as IVF or ICSI
* Has a phone that is known to be incompatible with COTS

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 1000 (Actual)
Dates: Start 2018-01-29 (Actual); Primary Completion 2018-09-19 (Actual); Study Completion 2018-09-19 (Actual)

PRIMARY OUTCOMES:
Difference in pregnancy rates across 2 cycles of use between volunteers trying to conceive in the home setting using (i) COTS, (ii) no intervention. | 2 months
  The difference in pregnancy rates between volunteers trying to conceive in the home setting using (i) COTS (ii) no intervention

SECONDARY OUTCOMES:
Assessment of behaviour of women trying to conceive | 2 months
  Quantitative assessment in methods used to try and help with conception and intercourse patterns.
Evaluation of women's experience of trying to conceive using COTS compared to not using ovulation tests | 2 months
  Qualitative interview responses regarding usage and experience of COTS or other methods whilst trying to conceive.

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Johnson, Dr, Study Director — SPD Development Company Ltd.
Locations (1):
- SPD Development Company Ltd, Bedford, Bedfordshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Johnson S, Bond S, Grace B, Marriott L. Increased Chance of Live Birth Following Use of Connected Ovulation Test System: Outcome Results from a Randomized Controlled Trial. Womens Health Rep (New Rochelle). 2022 Jan 31;3(1):60-66. doi: 10.1089/whr.2021.0102. eCollection 2022. PMID 35136878